CLINICAL TRIAL: NCT02325479
Title: Local Uterine Application of Low Molecular Weight Heparin (LMWH) in Intra-cytoplasmic Sperm Injection (ICSI) a Randomised Controlled Pilot Study
Brief Title: Local Uterine Application of Low Molecular Weight Heparin (LMWH) in Intra-cytoplasmic Sperm Injection (ICSI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Egyptian IVF-ET Center (Other)
Responsible Party: Principal Investigator, Mona Aboulghar, Professor Obstetrics and Gynecology Fetal Medicine unit Cairo University, IVF Consultant Egyptian IVF center -Maadi Cairo, The Egyptian IVF-ET Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 152014
Record Dates: First submitted 2014-12-17; First posted 2014-12-25 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: Low Molecular Weight (LMWH) Heparin ICSI Enaoxaprin sodium
MeSH Terms: conditions — Infertility | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): After scheduled oocyte pick up, a mock embryo transfer will be done using labotec catheter (Labotec, Gottingen Germany), and an injection of Enaoxaprin sodium (LMWH) (Clexane® Sanofi S.A Paris, France) will be given intrauterine in group A patients, 500 IU of LMWH which is 5mg, in 0.05 ml.
  Interventions: Drug: Enaoxaprin sodium
- Group B (Placebo Comparator): The control arm (group B) will be injected intrauterine with similar volume of tissue culture media (G.2 plus ref. 10132, Vitrolife)
  Interventions: Drug: tissue culture media

INTERVENTIONS:
Drug: Enaoxaprin sodium — intrauterine administration after oocyte pickup as the main experimental intervention
  Other Names: Clexane
  Arms: Group A
Drug: tissue culture media — intrauterine administration after oocyte pickup as placebo
  Other Names: (G.2 plus ref. 10132, Vitrolife)
  Arms: Group B

SUMMARY:
Heparin also has the ability to bind with and modulate a wide variety of proteins, which can influence a number of physiological processes involved in implantation & trophoblastic development. These processes include adhesion of the blastocyst to the endometrial surface & trophoblastic differentiation & invasion.

A recent Cochrane review hinted towards research to study the possible effects of the local (uterine), & NOT SYSTEMIC application of heparin during Assisted reproductive technology (ART). Based on the above evidence the investigators hypothesize that low molecular weight heparin given intrauterine at mock embryo transfer after oocyte pick up will help improve pregnancy rates in patients undergoing ART.

DETAILED DESCRIPTION:
Following ethical approval of the committee of Egyptian IVF-ET center, a pilot prospective randomized controlled study will include 40 patients, in which the study arm (group A ) will be injected with LMWH intrauterine during mock embryo transfer, just after ovum pickup, while the control arm (group B) will be injected intrauterine with similar volume tissue culture media (G.2 plus ref. 10132, Vitrolife) also after ovum pickup. Admission into either group will be through randomization after inclusion & exclusion criteria have been met and before start of controlled ovarian stimulation protocol.

The standard long gonadotrophin-releasing hormone (GnRH) agonist protocol will be used for patients with predicted normal response based on clinical & hormonal profile ; 1 mg of leuprolide acetate daily s.c injection (Lucrin ®; Abbott, Hoofddorp, The Netherlands) is applied from the mid luteal phase onward till the day of human chorionic gonadotropin (HCG) injection.

Gonadotropins in the form of human menopausal gonadotropin (HMG) (Merional ®, IBSA, Institut Biochimique SA, Lugano, Switzerland) will be given by intramuscular injection (IM) from the 2nd day of menstruation, The starting dose range from 150 to 450 IU depending on the basal follicle stimulating hormone (FSH) level, Antral follicle count (AFC) , Patient's age and body mass index (BMI).

In all protocols, stimulation is monitored by trans vaginal ultrasonography and serial estradiol (E2) measurements starting from day 7 of the cycle and the gonadotropin dose is adjusted individually according to follicular response.

After the development of at least three leading follicles≥18 mm, 10,000 unit of HCG (Choriomon, IBSA, Institut Biochimique SA) is given IM, and a trans-vaginal ultrasound-guided oocyte retrieval is performed 36 hours later.

After scheduled oocyte pick up, a mock embryo transfer will be done using labotec catheter (Labotec, Gottingen Germany), and an injection of Enaoxaprin sodium (LMWH) (Clexane® Sanofi S.A Paris, France) will be given intrauterine in group A patients.

LMWH is safe in pregnancy, category B drug , and given empirically sometimes in luteal phase and in early 1st trimester without reported problems, it has a half life of 4 Hours, and therefore it should not have any negative effects on developing embryos as it will not be present at the time of transfer while already performing it s desired effect on the endometrium.

The dose of LMWH given was calculated comparatively according to the work done by our group Mansour et.al, 2011, where intrauterine administration 500 IU of HCG improved the implantation and pregnancy rates.

Given the fact that this has not been attempted before, the best way to compare two different drugs is through biological activity. So if the investigators want to use 500 IU of LMWH, and knowing that In the in vitro purified system, enoxaparin sodium has a high anti Xa activity (approximately 100 IU/mg), so to get 500 IU of LMWH we need 5mg. Clexane 20mg is packed in a 0.2ml syringe, And therefore the investigators need to inject 0.05ml intrauterine using labotec catheter. (1/4 OF THE ORIGINAL SYRINGES CONTENT..i.e 5mg).

The control arm (group B) will be injected intrauterine with similar volume of tissue culture media (G.2 plus ref. 10132, Vitrolife) Oocytes are then fertilized in vitro using ICSI and after three to five days embryo transfer will be done using labotec catheter (Labotec, Gottingen Germany) with ultrasound guidance.

Progesterone pessaries 400 mg twice daily (Cyclogest 400mg ®Actavis plc. Dublin, Ireland) is given as a luteal support starting from the day of embryo transfer and continued for 16 days after.

Pregnancy is defined as the occurrence of a positive β-HCG >10 IU on day 12 after embryo transfer and a second higher value 2 days later, followed by ultrasonography confirmation of cardiac activity at 6 weeks gestation

A third party not involved in the actual study will moniter progress of the results and record them. Study will be stopped if more than 10 consecutive patients fail to get pregnant in the LMWH group. If the pregnancy rate >25% in the intervention group by the end of 20 cases, then recruitment willl continue till 60 patients are enrolled on each study arm.

ELIGIBILITY:
Inclusion Criteria:

1. Normal serum prolactin level & thyroid stimulating hormone (TSH)
2. Unexplained infertility
3. Tubal factor infertility
4. BMI <30 kg/m2

Exclusion Criteria:

1. Reduced ovarian reserve by AFC, Anti-mullerian hormone (AMH)
2. Presence of non disconnected hydrosalpinges
3. Frozen embryo transfer cycles
4. Uterine Anomalies
5. Submucous fibroids and polyps
6. Uterine synechia
7. Contraindication of pregnancy e.g.: Somatic and mental diseases, which are contraindications for carrying of a pregnancy and childbirth, inborn malformations or acquired deformations of uterus cavity which make embryo implantation or carrying of a pregnancy impossible ,ovarian tumors

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 14 days
  safety

SECONDARY OUTCOMES:
Early miscarriage rate | 12 weeks
Implanation rate | 3 weeks after ET

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Aboulghar, M.D, Principal Investigator — IVF consultant
Locations (1):
- The Egyptian IVF-ET Center, Cairo, Maadi, Egypt

REFERENCES:
- [Background] Akhtar MA, Sur S, Raine-Fenning N, Jayaprakasan K, Thornton J, Quenby S, Marjoribanks J. Heparin for assisted reproduction: summary of a Cochrane review. Fertil Steril. 2015 Jan;103(1):33-4. doi: 10.1016/j.fertnstert.2014.09.005. Epub 2014 Oct 1. PMID 25282470
- [Background] Mansour R, Tawab N, Kamal O, El-Faissal Y, Serour A, Aboulghar M, Serour G. Intrauterine injection of human chorionic gonadotropin before embryo transfer significantly improves the implantation and pregnancy rates in in vitro fertilization/intracytoplasmic sperm injection: a prospective randomized study. Fertil Steril. 2011 Dec;96(6):1370-1374.e1. doi: 10.1016/j.fertnstert.2011.09.044. Epub 2011 Nov 1. PMID 22047664